CLINICAL TRIAL: NCT06287996
Title: Chief Nursing Officer, Nursing Department, Mackay Memorial Hospital
Brief Title: Effects of Warm Water Footbath Intervention on Sleep Quality , Fatigue and Heart Rate Variability in Patients With Heart Failure
Status: Enrolling by invitation | Phase: Not Applicable | Type: Interventional
Sponsor: Mackay Memorial Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 23MMHIS503e NA
Record Dates: First submitted 2024-02-24; First posted 2024-03-01 (Actual); Last update posted 2024-03-01 (Actual); Status verified 2024-02

CONDITIONS: Footbath; Heart Failure; Sleep Quality; Fatigue; Heart Rate Variability
MeSH Terms: conditions — Heart Failure; Sleep Initiation and Maintenance Disorders; Fatigue | interventions — Actigraphy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Warm water foot-bath and actigraphy (Experimental): Warm water foot-bath and actigraphy
  Interventions: Other: footbath and actigraphy; Device: actigraphy
- actigraphy (Active Comparator): actigraphy
  Interventions: Device: actigraphy

INTERVENTIONS:
Other: footbath and actigraphy — Receive warm water foot bath for 4 weeks, 1 hour before going to bed every night (7-9PM), temperature 42℃ for 20 minutes, water depth 10cm above the ankle joint and wearing an actigraphy for 4 weeks
  Arms: Warm water foot-bath and actigraphy
Device: actigraphy — Wearing an actigraphy for 4 weeks

SUMMARY:
This study adopted an experimental research design to explore the effects of a warm water foot bath program on fatigue, sleep, and heart rate variability in patients with heart failure. The subjects of the study were heart failure patients in the cardiology outpatient department. The patients were randomly assigned to the experimental group and the control group. The control group received routine care and wore an actigraph. The experimental group received 4 additional care in addition to routine care and wearing an actigraph. Weekly warm water foot bath, data collection includes subjective sleep quality and fatigue level, physiological measurements: sleep quality-sleep time and efficiency, and heart rate variability index.

DETAILED DESCRIPTION:
This study adopted an experimental research design to explore the effects of a warm water foot bath program on fatigue, sleep, and heart rate variability in patients with heart failure. The research subjects are cardiology outpatients at two medical centers in northern China (Taipei and New Taipei City). It is expected to recruit 76 research subjects (38 in the control group and 38 in the experimental group). Pre-test data collection includes basic personal information, subjective sleep quality and fatigue level questionnaires, and wearing an actigraph on the wrist. Patients were assigned to an experimental group and a control group based on random assignment results. The control group received routine care and wore an actigraph. In addition to routine care and wearing an actigraph, the experimental group also received warm foot baths for 4 weeks, one hour before going to bed every night. (7-9PM), the temperature is 42°C for 20 minutes, and the water depth is 10 cm above the ankle joint. Both groups receive weekly phone calls to confirm wearing the actigraph and performing warm water foot baths. Post-test data were collected in the second and fourth weeks, including subjective sleep quality and fatigue level questionnaires. After the four weeks, the researchers collected and analyzed physiological measurements: sleep quality-sleep time and efficiency, and heart rate variability index. Research tools include basic information sheets, actigraphy, warm water foot bath machines, Pittsburgh Sleep Quality Scale, and Piper Fatigue Scale. The collected data were processed and analyzed using SPSS 26.0 statistical software. Warm water foot bath is a local hot compress, which is non-invasive and simple to operate. It has the effect of relieving sleep and fatigue of patients with heart failure. It is suitable for patients with heart failure during hospitalization or at home.We hope it will be helpful to clinical care practice, education and research.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosed by a cardiologist as suffering from heart failure, NYHA functional class one to three and with a history of reduced ejection fraction (HFrEF, EF ≤ 40%)
* Clear consciousness and able to communicate
* Those who can maintain a sitting position by themselves or with the help of others
* Temperature, hearing and vision are normal

Exclusion Criteria:

* Leg injury or foot wound
* Peripheral vascular disease
* History of stroke

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 76 (Estimated)
Dates: Start 2024-02-23 (Estimated); Primary Completion 2024-06-01 (Estimated); Study Completion 2024-08-01 (Estimated)

PRIMARY OUTCOMES:
sleep quality | Before intervention and the 2nd and 4th week after intervention

SECONDARY OUTCOMES:
fatigue | Before intervention and the 2nd and 4th week after intervention

OTHER OUTCOMES:
heart rate variability | Fourth week after intervention

CONTACTS AND LOCATIONS:
Locations (1):
- Mackay Memorial Hospital, Taipei, Zhongshan, Taiwan

IPD SHARING:
Plan to Share IPD: No